CLINICAL TRIAL: NCT03259256
Title: Islet Allotransplantation for Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-03
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic transplantation of human islet (Experimental): Each subject may receive 1-3 transplantations of allogeneic human islets we will inject the least dose of 3,000 IEQ/kg body weight of the recipient. Tacrolimus 1 mg p.o. bid adjusted to reach target trough levels of 3-6 ng/ml.
  Interventions: Procedure: Allogeneic transplantation of intrahepatic islet

INTERVENTIONS:
Procedure: Allogeneic transplantation of intrahepatic islet — Allogeneic transplantation of intrahepatic islet is one of the effective methods for diabetic therapy

SUMMARY:
The purpose of this study is to determine if islet cell transplantation , is an effective treatment for type 1 diabetes. Study participants may receive up to three islet transplants and will be followed for five years to monitor blood sugar control, islet transplant function, and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of type 1 diabetes 18 <Age <70 years Evolution of diabetes for more than 5 years Regular patient follow-up (> or equal to 2 visits per year from the same diabetologist) ABO compatibility with the donor Cross match negative Anti-HLA antibodies (class I and / or class II) detected by lymphocytotoxicity <20% Accepting patients effective contraception during the study period

Exclusion Criteria:

Clinical diagnosis of type 2 diabetes BMI > 28 Need insulin < 28 U per day Pregnancy, lactation Psychiatric Disorders Inability to communicate or cooperate with the investigator Lack of therapeutic compliance, including HbA1C > 12% Chronic liver disease Proliferative retinopathy unstabilized History of cancer, whatever the date, except for basal or squamous cell skin cancers over 1 year.

Systemic infection Chronic high risk of requiring corticosteroids Need for long-term corticosteroid, outside that specified in renal transplantation, the patients will be weaned before transplantation Anticoagulant vitamin K or antiplatelet treatments Platelets < 100 giga/L and/or neutrophils <1.5 giga/L Chronic intoxication by alcohol, tobacco, or other substance (abstinence > 6 months required) Active infection by hepatitis B, hepatitis C and HIV, HTLV-1-HTLV2 Ascites

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-04-23 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Obtaining an improvement in glycemic control | nine months after first and last islet transplants
  The proportion of subjects with an HbA1c ≤ 6.5% and free of severe hypoglycemic events
normal glycemic control without insulin | 3 months after graf
  A fasting glucose (> 8 hours) less than 1.25 g/L and a 2 hours glucose after oral intake of 75g of glucose, less than 2 g/L in a patient without insulin for at least 15 consecutive days during the the first 6 months

SECONDARY OUTCOMES:
insulin independence | One year after the last transplant
  insulin independence
Hypoglycemic episodes by HYPO score | 3 months after transplantation
  Hypoglycemic episodes by HYPO score
degenerative complications of diabetes | 18 months after transplantation
  degenerative complications of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: ping Xue, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No